CLINICAL TRIAL: NCT05691530
Title: Phase 1 Trial to Model Primary, Secondary, and Tertiary Dengue Using a Monovalent Vaccine
Brief Title: Trial to Model Primary, Secondary, and Tertiary Dengue Using a Monovalent Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10001078; 001078-I
Record Dates: First submitted 2023-01-19; First posted 2023-01-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10-01

CONDITIONS: Response To Dengue Exposure
Keywords: Viremia; Geometric Mean Titer; Safety; Immunogenicity; Sequential Exposure; Lymph Node Aspirates
MeSH Terms: conditions — Viremia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Flavivirus Naive (Experimental): Those with <=50% neutralization at a 1:10 dilution to all four DENV serotypes, no history of flavivirus vaccination, or travel history that increases the likelihood of other flavivirus infections.
  Interventions: Drug: rDENdelta30/31-7164
- Polytypic DENV Antibody Profile (Experimental): Those considered immune (a >=70% neutralization or plaques at a 1:40 dilution) to at least two serotypes.
  Interventions: Drug: rDENdelta30/31-7164
- Primary Heterotypic DENV Antibody Profile (Experimental): Those who have a >=70% neutralization or plaques at a 1:40 dilution for a single serotype, either DENV1, DENV2, or DENV4.
  Interventions: Drug: rDENdelta30/31-7164

INTERVENTIONS:
Drug: rDENdelta30/31-7164 — The rDEN3delta30/31-7164 vaccine is a live attenuated virus constructed by creating two deletions in the 3 UTR of the DENV3 Sleman/78 strain. The rDEN3delta30/31-7164 vaccine will be delivered subcutaneously into the left deltoid area on day 0. The vaccine dose will consist of 0.5 mL of 10^3 PFU/mL of rDEN3delta30/31-7164 plus Plasma-Lyte A pH 7.4 diluent.

SUMMARY:
Background:

Dengue is a disease caused by a virus transmitted by mosquitoes in tropical and subtropical regions. Dengue is a leading cause of hospital stays and death in parts of Asia and Latin America, and outbreaks have occurred in the US. Currently, only one vaccine is licensed for dengue, but it only protects people who have had dengue before. In people who have never had dengue, that vaccine increases the risk of severe disease. Better vaccines are needed.

Objectives:

To test a potential new vaccine against dengue. To see if side effects and immune responses are different depending on a person s previous exposure to dengue.

Eligibility: Healthy people aged 18 to 59 years.

Design:

Participants will visit the clinic 11 times in 7 months; 9 of those visits will be in the first 2 months. Two additional visits are optional.

Participants will be screened. They will have a physical exam with urine and blood tests. They will complete a survey about their travel history.

Participants may opt to have a lymph node aspiration before receiving the study vaccine. An area in the left armpit will be numbed. A needle will be inserted to remove some cells from a lymph node.

The vaccine will be injected into the fat under the skin of the participant s upper left arm.

Participants will return for a provider visit and blood draws every 3 days for about the first 2 weeks. Then they will return for a provider visit and blood draws after longer intervals up to 7 months. The lymph node aspiration may be repeated at later visits.

Participants may opt to return for a last visit after 12 months.

DETAILED DESCRIPTION:
Study Description:

Phase 1 trial wherein healthy adults with no (naive), one (primary heterotypic), or more than one (polytypic) previous natural dengue virus (DENV) infection(s) will be immunized with the DENV3 monovalent vaccine rDEN3delta30/31-7164. We aim to examine how pre-vaccine host immunity influences the safety and immunogenicity of monovalent DENV3 vaccination in a non-endemic population. We hypothesize that the vaccine will be safe and well tolerated, and all groups will have evidence of infection with the vaccine strain as indicated by a significant increase in the DENV neutralizing antibody geometric mean titer (GMT) between days 0 and 28. However, due to the immunity conferred by prior dengue exposure(s), the polytypic group will have the lowest and the heterotypic group will have the highest mean peak viremia, indicating protection and enhancement, respectively. Additionally, the polytypic group will have the strongest CD8+ T-cell responses at day 15 and will only have a transient rise in GMT with no difference in GMT between days 0 and 57. In contrast, the change in GMT will persist at day 57 in the heterotypic and naive groups. Finally, we expect that prior immunity will influence the vaccine response as evidenced by a significant association between the day 0 GMT and GMT at days 28 and 57.

Primary Objective:

Evaluate the safety of monovalent DENV3 vaccination in those with distinct natural DENV infection histories living in non-endemic areas, and how prior DENV immunity influences protection against vaccine strain infection evaluated by the change in GMT and mean peak viremia.

Secondary Objective:

Further evaluate how DENV infection history impacts the immunogenicity of the vaccine.

Primary Endpoints:

1. The frequency and severity of local and systemic reactogenicity signs and symptoms during the 28-day period after each vaccination, unexpected adverse events (AEs) up to 28 days after each vaccination, and serious adverse events (SAEs) through day 180.
2. Change in DENV neutralizing antibody GMT between days 0 and 28.
3. Mean peak viremia among groups as measured by viral quantitative reverse transcription polymerase chain reaction (qRT-PCR) between days 3 and 15.

Secondary Endpoints:

1. Change in DENV neutralizing antibody GMT between days 0 and 57.
2. DENV neutralizing antibody GMT at days 0, 28, and 57.
3. Magnitude of the CD8+ T-cell response at day 15 among groups as measured by activation-induced marker (AIM) assays.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Aged 18 to 59 years.
* In good general health as evidenced by medical history, physical examination, and laboratory screening results.
* Willing to allow storage of samples and data for future research.
* Willing to forgo receipt of any vaccine in the 28 days preceding the vaccine or in the 28 days following the dose of vaccine. For participants opting for LN FNA on day 57, they must be willing to forgo any vaccine through final LN FNA.
* For individuals who can become pregnant: use of at least one method of highly effective contraception from the invitation to participate in the trial through day 60 after vaccination.
* Able to provide informed consent.
* Willing to adhere to lifestyle considerations for the duration of the study.
* Willing to avoid travel to a dengue-endemic area as defined by the Centers for Disease Control and Prevention (CDC) from 1 month before vaccination through day 57
* Baseline absolute neutrophil count (ANC) > 750 cells/microL.
* Baseline creatinine < 1.5 mg/dL.
* Baseline ALT < 1.25 (SqrRoot) upper limit of normal.
* Serologic evidence of previous dengue virus infection indicative of either one previous DENV1, 2, or 4 infection or infection with at least two different serotypes.

  --For the flavivirus-na(SqrRoot) ve group, they must have no history of flavivirus vaccination, medical illness concerning for a flavivirus infection, or travel history that increases the likelihood of other flavivirus infections. If there is uncertainty about a previous flavivirus exposure, then confirmatory antibody testing against the virus of interest must be negative.
* Agree to avoid participation in other clinical studies requiring investigational interventions for the duration of this study (180 days).
* Agree to avoid blood and plasma donation outside this study through day 28.

Contraceptive requirements: Participants who can get pregnant must agree to use highly effective contraception as outlined below from the invitation to participate in the study (approximately 2 weeks after screening) through day 60. Day 0 will be scheduled at least 28 days after the initiation of effective contraception. Participants who can get pregnant must have a negative pregnancy test on day 0 before receiving rDEN3DELTA30/31-7164. If a participant becomes pregnant or suspects they are pregnant by day 60, then they should inform the study staff and their primary care physician immediately. Acceptable forms of contraception are:

* Intrauterine device or equivalent.
* Hormonal contraceptive (eg, consistent, timely, and continuous use of contraceptive pill, patch, ring, implant, or injection that has reached full efficacy prior to dosing).
* Condom, diaphragm, or cervical cap plus spermicide.
* A stable, long-term monogamous relationship with a partner who does not pose any potential pregnancy risk, eg, has undergone a vasectomy at least 6 months prior to vaccination or is of the same sex as the participant.
* A hysterectomy and/or a bilateral tubal ligation, bilateral oophorectomy, or post-menopausal status defined as age >=45 years and at least 1 year since last menstrual period.

Pregnancy after day 60 will not be exclusionary as this will not impact our primary or secondary endpoints. Although we may observe pregnancy-associated differences in the transcriptome, these endpoints are exploratory and we have chosen to prioritize safety and inclusivity for people who can become pregnant. Study blood draw volumes after day 28 are less than the recommended volumes for research blood in critically ill patients. Pregnant participants will be excluded from LN FNA due to the potential risks of anesthetics that may be used. Pregnancy testing will be performed on each LN FNA day, with a negative result required to proceed to aspiration.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnant at screening.
* History of or positive test result for HIV, hepatitis B, or hepatitis C.
* History of previous dengue vaccine.
* Has any of the following:

  * More than 10 days of systemic immunosuppressive medications (>=10 mg prednisone dose or its equivalent) or cytotoxic medication within the 30 days prior to vaccination or immunomodulating therapy within 180 days prior to vaccination.
  * Received blood products, including immunoglobulin products, within 120 days prior to vaccination.
  * History of serious reactions to vaccines.
  * Hereditary, acquired, or idiopathic forms of angioedema.
  * Idiopathic urticaria within the past year.
  * Asthma that is not well controlled or required emergency care, urgent care, hospitalization, or intubation during the past two years or that requires the use of oral or intravenous steroids.
  * Type 1 or type 2 diabetes mellitus that is not well controlled (hemoglobin A1c > 8).
  * Clinically significant autoimmune disease or immunodeficiency.
  * Blood pressure >= 180/110 (stage 3 hypertension) on at least 2 measures.
  * Documented diagnosis of a bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
  * Significant bruising or bleeding difficulties with subcutaneous injections or blood draws.
  * Malignancy that is active or treated malignancy for which there is no reasonable assurance of sustained cure, or malignancy that is likely to recur during the study period.
  * Asplenia or functional asplenia.
  * Current alcohol or drug abuse or addiction and/or positive drug screen with substances other than marijuana.
* Any medical, psychiatric, or social condition that, in the judgement of the investigator, is a contraindication to protocol participation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in the DENV neutralizing antibody GMT between days 0 and 28. | Days 0 and 28
  Evaluate the safety of monovalent DENV3 vaccination in those with distinct natural DENV infection histories living in non-endemic areas, and how prior DENV immunity influences protection against vaccine strain infection evaluated by the change in GMT and mean peak viremia.
The frequency and severity of local and systemic reactogenicity signs and symptoms during the 28 day period after each vaccination, unexpected AEs up to 28 days after each vaccination, and SAEs through day 180. | Days 28 and 180
  Evaluate the safety of monovalent DENV3 vaccination in those with distinct natural DENV infection histories living in non-endemic areas, and how prior DENV immunity influences protection against vaccine strain infection evaluated by the change in GMT and mean peak viremia.
Mean peak viremia among groups as measured by viral qRT-PCR between days 3 and 15. | Days 3, 6, 9, 12 and 15
  Evaluate the safety of monovalent DENV3 vaccination in those with distinct natural DENV infection histories living in non-endemic areas, and how prior DENV immunity influences protection against vaccine strain infection evaluated by the change in GMT and mean peak viremia.

SECONDARY OUTCOMES:
Change in DENV neutralizing antibody GMT between days 0 and 57 and days 0 and 90. | Days 0, 57 and 90
  Further evaluate how DENV infection history impacts the immunogenicity of the vaccine.
DENV neutralizing antibody GMT at days 0, 28, 57, and 90. | Days 0, 28, 57 and 90
  Further evaluate how DENV infection history impacts the immunogenicity of the vaccine.
Change in DENV3 neutralizing antibody titer between day 0 and peak titer (measured at days 28, 57, or 90). | Days 0, 28, 57 and 90
  Further evaluate how DENV infection history impacts the immunogenicity of the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Camila D Odio, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Odio CD, Lowman KE, Law M, Aogo RA, Hunsberger S, Wood BJ, Kassin M, Levy E, Callier V, Firdous S, Hasund CM, Voirin C, Kattappuram R, Yek C, Manning J, Durbin A, Whitehead SS, Katzelnick LC. Phase 1 trial to model primary, secondary, and tertiary dengue using a monovalent vaccine. BMC Infect Dis. 2023 May 23;23(1):345. doi: 10.1186/s12879-023-08299-5. PMID 37221466
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001078-I.html